CLINICAL TRIAL: NCT03775694
Title: Diffusion MRI-1 Imaging Database
Acronym: dMRI-1
Status: Completed | Type: Observational
Sponsor: Medtronic Spinal and Biologics (Industry)
Responsible Party: Sponsor
Other Study IDs: MDT17084
Record Dates: First submitted 2018-12-12; First posted 2018-12-14 (Actual); Last update posted 2022-05-04 (Actual); Status verified 2022-05

CONDITIONS: Epilepsy; Tumor; Healthy; Other
MeSH Terms: conditions — Epilepsy; Neoplasms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

INTERVENTIONS:
Device: dMRI Scan — Data will be collected from cases where dMRI scans were obtained as part of the subject's previous treatment.

SUMMARY:
The purpose of the dMRI-1 data collection study is to establish a database of clinical images and limited medical history information from patients that have previously received a dMRI scan. All data collected will be de-identified. No safety or effectiveness assessments will be completed.

ELIGIBILITY:
Inclusion Criteria:

1. Patient is either ≥ 18 years and has previously received an acceptable dMRI scan(s) with at least 30 unique gradient directions or < 18 years who has previously received an acceptable dMRI scan of any number of unique gradient directions and who is allowed to participate in this type of research project (e.g., IRB/EC approval with waiver of consent) per IRB/EC
2. Acceptable dMRI scan was completed prior to site activation in the study

Exclusion Criteria:

None

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Patients who have previously received a dMRI scan.
Sampling Method: Non-Probability Sample
Enrollment: 299 (Actual)
Dates: Start 2019-06-06 (Actual); Primary Completion 2022-04-29 (Actual); Study Completion 2022-04-29 (Actual)

PRIMARY OUTCOMES:
Image assessment | Procedure

CONTACTS AND LOCATIONS:
Locations (6):
- United States (3):
  - University of Colorado, Aurora, Colorado
  - University of Florida, Gainesville, Florida
  - Seattle Children's Hospital, Seattle, Washington
- Canada (3):
  - University of Calgary, Calgary, Alberta
  - The Hospital for Sick Children, Toronto, Ontario
  - University of Sherbrooke, Sherbrooke, Quebec